CLINICAL TRIAL: NCT03464812
Title: Evaluating Patient Engagement and Other Outcomes for Ethnically Diverse Patients With Type 2 Diabetes Participating in a Structured, Physician Supported, Patient-centered Diabetes Education Program
Brief Title: Evaluating Outcomes for Ethnically Diverse Patients With Type 2 Diabetes Participating in a Diabetes Education Program
Acronym: DSMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RADC2018_1
Record Dates: First submitted 2018-03-02; First posted 2018-03-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-08

CONDITIONS: Type2 Diabetes
Keywords: Diabetes education; Psychosocial management of diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DSMES Group (Other): Patients with type 2 diabetes will undergo a diabetes education program (DSMES) and evaluated for outcomes before and after completing the program.
  Interventions: Behavioral: DSMES

INTERVENTIONS:
Behavioral: DSMES — It is primarily an educational intervention that is focused on assisting patients improve their management and coping with type 2 diabetes.

SUMMARY:
The proposed study has been developed to evaluate patient, physician, and provider (educator) centered barriers to and facilitators for engaging in the Diabetes Self Management Education and Support (DSMES) and developing a patient-centered, physician supported DSMES program that could potentially address barriers shared by the patients and their healthcare professionals (Phase 1). The feasibility and efficacy of the newly developed program will be evaluated with an ethnically diverse cohort of 90 patients with type 2 diabetes (30 Caucasians, Asians, and Hispanics each) (Phase 2). A variety of outcomes including clinical, behavioral and psycho-social measures will be used to assess program acceptability and effectiveness.

DETAILED DESCRIPTION:
Diabetes is a chronic and a progressive metabolic disorder which necessitates active patient involvement to effectively manage nutrition, physical activity, and medication for optimal outcomes. Self-management is a critical aspect of diabetes care and a variety of studies have established the need for people with diabetes to be knowledgeable about their condition and be actively involved in its management to effectively reduce the risk of future health complications and improve other outcomes. Diabetes self-management education and support (DSMES) can help patients effectively engage in and perform their diabetes-related self-care activities. However, only a small number of patients with diabetes participate in DSMES. A few studies in this area have highlighted both physician and patient-related factors that could affect the receipt of DSMES. Patients' involvement in a DSMES program continues to be largely prompted by a physician referral and it has been suggested that improving physician involvement in the DSMES process could enhance overall patient engagement and adherence to such programs.

As part of the proposed mixed methods study, in Phase 1, in-depth surveys (or interviews) will be undertaken with: (a) physicians caring for people with type 2 diabetes, (b) DSMES providers (e.g., certified diabetes educators, diabetes nurses, dietitians), and (b) patients with type 2 diabetes regarding their perception of diabetes education programs, barriers, and facilitators to engagement. Findings from Phase 1 will be shared with the education team at a diabetes center in a community hospital in Orange County, California to inform changes to their currently existing diabetes education curriculum to make it more patient-centered and improve physician engagement and support. As part of Phase 2, the newly developed program will be implemented with a diverse cohort of 90 patients with type 2 diabetes. Patient participation (attendance) in the DSMES process will be documented as a primary marker of patient engagement while their clinical and psycho-social outcomes will serve as secondary indicators. Among other outcomes, physician, educator, and patient satisfaction with the newly developed referral process will also be assessed as a measure of intervention acceptability and success.

ELIGIBILITY:
Inclusion Criteria:

Patients of White, Asian, or Hispanic origin (30 in each group) Fluent in English (for the White and Asian group) Fluent in Spanish (for the Hispanic group) Age > 18 years Physician referral for DSME/S Formal diagnosis of type 2 diabetes

Exclusion Criteria:

Current or planned pregnancy. Any medical or other condition that the investigator feels would interfere with study participation.

Mental incapacity precluding adequate understanding or cooperation. Potential participants who are imprisoned or hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Program completion | Approximately at 4 months from the start of the study.
  Evaluate the rate of program completion in study participants

SECONDARY OUTCOMES:
Glycemic control | At baseline and repeated after approximately 4 months
  Evaluated using HbA1c (blood test)
Diabetes-specific quality of life | At baseline and repeated after approximately 4 months
  Measure assessing diabetes-specific quality of life
Diabetes-related distress | At baseline and repeated after approximately 4 months
  Measure assessing diabetes-related distress or problem areas in diabetes
Diabetes self-care | At baseline and repeated after approximately 4 months
  Measure assessing diabetes-related self-care
Diabetes-related self efficacy | At baseline and repeated after approximately 4 months
  Measure assessing diabetes-related self-efficacy
Patient and referring provider satisfaction | Approximately at 4 months from the start of the study.
  Measures to assess patient and referring provider related satisfaction with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Harsimran Harsimran, PhD, Principal Investigator — Hoag Hospital
Locations (1):
- Mary & Dick Allen Diabetes Center, Hoag Hospital, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No